CLINICAL TRIAL: NCT01249625
Title: Incidence of Respiratory Illness in Outpatient Healthcare Workers Who Wear Respirators or Medical Masks While Caring for Patients
Brief Title: The Respiratory Protection Effectiveness Clinical Trial
Acronym: ResPECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); US Department of Veterans Affairs (U.S. Federal Agency); University of Massachusetts, Amherst (Other); Denver Health and Hospital Authority (Other); Children's Hospital Colorado (Other); VA Eastern Colorado Health Care System (U.S. Federal Agency); VA New York Harbor Healthcare System (U.S. Federal Agency); Michael E. DeBakey VA Medical Center (U.S. Federal Agency); Washington D.C. Veterans Affairs Medical Center (U.S. Federal Agency); VA St. Louis Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: NA_00031266
Record Dates: First submitted 2010-11-29; First posted 2010-11-30 (Estimated); Results first posted 2019-04-25 (Actual); Last update posted 2019-04-25 (Actual); Status verified 2019-04

CONDITIONS: Influenza; Respiratory Syncytial Viruses; Paramyxoviridae Infections; Coronavirus; Rhinovirus
Keywords: Influenza; H1N1; Respiratory protection; N95 respirator; Medical mask; Personal protective equipment; Facial protective equipment; Pandemic planning
MeSH Terms: conditions — Influenza, Human; Paramyxoviridae Infections; Coronavirus Infections | interventions — N95 Respirators; Peak Expiratory Flow Rate

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- N95 Respirator (Active Comparator): The investigators are comparing specific N95 respirator against specific medical masks.
  Interventions: Device: N95 Respirator
- Medical/surgical mask (Active Comparator): The investigators are comparing medical/surgical masks against the N95 respirator.
  Interventions: Device: Medical/surgical mask

INTERVENTIONS:
Device: N95 Respirator — Participants in this arm will be asked to wear an N95 respirator for the extent of the 12 week study period.
  Other Names: 3M Corporation 1860, 1860S, and 1870 models; Kimberly Clark Technol Fluidshield Particulate Filter Respirator (PFR) 95-170; PFR 95-174
  Arms: N95 Respirator
Device: Medical/surgical mask — Participants in this arm will be asked to wear a medical/surgical mask for the extent of the 12 week study period.
  Other Names: Precept 15320; Kimberly Clark Technol Fluidshield 47107
  Arms: Medical/surgical mask

SUMMARY:
Despite widespread use of respiratory protective equipment in the U.S. healthcare workplace, there is very little clinical evidence that respirators prevent healthcare personnel (HCP) from airborne infectious diseases. Scientific investigation of this issue has been quite complicated, primarily because the use of respirators has become "the standard of care" for protection against airborne diseases in some instances, even without sufficient evidence to support their use. The key question remains: How well do respirators prevent airborne infectious diseases? The answer to this important question has important medical, public health, political and economic implications.

DETAILED DESCRIPTION:
Prevention strategies are key in limiting the transmission of respiratory viruses such as influenza. Among non-pharmacologic interventions, there is intense interest in the use of facial protective equipment (FPE) - medical masks (MM) or N95 respirators (N95) - as a key component of personal protective equipment (PPE) when faced with respiratory illness including influenza. However, their relative protective effect is unknown, especially in the outpatient setting (OPD). To plan for future epidemics and best manage limited supplies of FPE, evidence is needed to guide planning activities and policy makers. This project aims to answer a key question: How do N95s protect healthcare workers (HCWs) in the OPD against influenza, influenza-like illness (ILI), acute respiratory illness (ARI) and other causes of respiratory illnesses including respiratory viral illness (RV), as compared to MMs? The study outcomes are to:

* determine the most effective FPE equipment to use to prevent disease transmission in the OPD during an influenza outbreak, epidemic or pandemic event.
* the incidence of organism-specific rates of ARI in the OPD during the RV season.
* the incidence rate of organism-specific respiratory viral infections in the OPD.

Clinics (or their functional partitions) will be randomized into either the N95 or MM arm using a stratified randomization scheme to ensure comparability between the two arms. All participants, regardless of study arm, will be fit-tested for an N95. The study will require a 16-18 week period that will be initiated when viral surveillance data indicates that influenza season has begun. Participants will be recruited through informational meetings with clinic staff. Participants will have blood drawn before week 1 and after the end of the active portion of the study to assess seroconversion over the study period to capture the incidence of non-symptomatic influenza. All participants will fill out a pre-study survey and post on knowledge, attitudes and beliefs regarding influenza, influenza vaccinations, and appropriate PPE.

During the first week, participants will fill out a form with basic demographic and workplace information. Participants will be asked to 1. wear participant's appropriate FPE when in close contact with patients with suspected or confirmed influenza or RV for the next 12-16 weeks; 2. fill out a daily form assessing exposure to ILI and FPE use, and weekly forms assessing RV symptoms and medication use. The investigators will collect nasal and throat (pharyngeal) swabs twice during the study for all participants, and when participants report having an ILI or ARI. Study staff will make unannounced visits to the clinics to observe FPE and hand hygiene compliance rates.

Participants will be compensated for participation (as detailed below). To be included the clinical site leadership has agreed to have one of more participants in the trial. To be included the subject(s): (1) meets the definition of "healthcare personnel" (2) is able to read and sign informed consent (3) agrees to all requirements of the protocol, including fit testing and diary keeping (4) is 18 years old or greater (6) passes fit testing for one of the study supplied N95 and agrees to use that model for the entire 16 week period of the study. Subjects are excluded if: (1) subject self-identified as having severe heart, lung, neurological or other systemic disease that one or more Investigator believes could preclude safe participation (2) are known to not tolerate wearing FPE for any period (3) facial hair, or other issue such as facial adornments, preclude respirator Occupational Safety and Health Administration (OSHA)-compliant fit testing or proper mask fit during the study period (4) subjects are advised by Occupational Health (or other qualified clinician) to not wear the same or similar respirator or medical mask models used in this study (5) in the opinion of the Investigator, may not be able to reasonably participate in the trial for any reason (6) Self-identified as in, or will be in the third trimester of pregnancy, during the study period.

Participants will be compensated for participation. Due to space limitations details are not presented here but are available from the overall study PI's.

During the study period, study staff will be making unannounced visits to the clinics to measure hand hygiene and FPE compliance. The information collected will not be shared with the supervisors or administration of the clinics.

Respiratory Protection Effectiveness Clinical Trial (ResPECT) Analysis Plan

1. Analysis timeline and procedures

   A pre-specified analysis plan for the primary manuscript of ResPECT was initially approved by all study principal and study-site lead investigators on April 2016 and updated in May 2017 to reflect the addition of the Laboratory Detected Respiratory Infection (LDRI) outcome to the analysis. At the time of this revision (a) all data collection is complete, (b) all laboratory specimen samples have been tested for the primary and secondary outcomes, and (c) the database housing all of the ResPECT data contained no information about which clinics were assigned to which arm of the study. Once the analysis plan is updated and changes submitted to the site IRB's, the data coordinating center will release labels that identify separate arms of the study to the ResPECT statisticians who will use those codes to implement the analysis as described in this document.
2. General outline of analysis framework

The ResPECT study was a cluster-randomized trial that used constrained randomization (i.e. matching) to ensure balance across arms. The analysis described in this document is an unmatched analysis, i.e. the analysis does not explicitly account for the matching. This has been described as an appropriate approach to analyzing data arising from a matched design.

The final analysis of ResPECT outcome data will consist of intention-to-treat (ITT) and per-protocol analyses (PP) for each of the five study outcomes defined below. For each analysis, the investigators will fit and report results from both adjusted and unadjusted models. Unadjusted models will be analyzed at the cluster-level, and will only include a main effect estimate for the mask and the cluster-level random effects to account for repeated measures of related clusters across multiple seasons. Adjusted models will be analyzed at the individual-level and will include individual-level covariates and random effects to account for repeated measures of the same individual across seasons.

2.a Intention-to-treat analysis The ITT analysis will include all of the ResPECT participants who were randomized- i.e., those assigned a mask based on participant's clinic affiliation. Participant's data will be included according to participant's treatment assignment, regardless of participant's adherence to protocol, subsequent withdrawal, failure to provide requested data/samples, or loss to follow-up. This analysis is intended to capture a more realistic outcome of intervention by acknowledging that noncompliance and protocol deviations are an unavoidable part of clinical practice.

In this study, any person who was eligible according to the baseline survey will be included in the ITT analysis. The outcomes for many participants will be missing, particularly those who withdrew during the course of the study. This missingness could conceivably be (a) related to outcome/illness status if individuals were more likely to quit the study because the individuals became sick, or (b) related to the assigned intervention if those assigned one mask over another were more likely to withdraw from study participation. The investigators will assess possible relationships between self-reported reasons for withdrawal and measured variables. Approaches for imputing missing data are addressed below.

2.b Per-protocol analysis Any participant who completed at least eight weeks of study participation will be included in the per protocol analysis. This strategy will include some participants who only had one blood draw or who are missing reliable serological data due to timing of or lack of information on vaccination (see Participant flow for ResPECT study analysis approaches showing ITT and per protocol cohorts and Decision Algorithm for serological influenza outcome adjudication below). These inclusion/exclusion criteria were decided on by the study PIs.

The reasons for missing participant blood samples include loss to follow-up with or without formal withdrawal/deactivation, sample loss due to handling/labeling error, or insufficient sample volume. Since the serologic definition of influenza seroconversion is a 4-fold increase in titer, unpaired serology cannot be assigned an influenza seroconversion status and must be imputed. Missing serologic data will not exclude the patient from the polymerase chain reaction (PCR)-laboratory assessment. Hence, if an individual is missing a second blood draw but had lab-confirmed influenza by PCR, then this individual will be considered to have had a lab-confirmed influenza outcome. This may create non-random missingness, but it was decided by PIs that since this would not impact many study participants the risk of bias to the overall study was very low.

2.c Handling of missing data via imputation methods There will be substantial missing data in the outcome (lab-confirmed influenza) and other covariates. The missing data will be imputed using standard multiple imputation techniques, creating imputed datasets with no missing values for each analysis. Each of these datasets will be analyzed using the regression models described below. The results from all of the analyses will be pooled using standard multiple imputation techniques for combining estimates across imputed datasets.

2. d Process for determining participant membership in ITT and per protocol cohorts Participants signed informed consent. Those who failed to meet inclusion criteria or did not complete screening were excluded. Those who met the inclusion criteria were randomly assigned to a mask group and formulate the ITT cohort. The 'per protocol' cohort will not include those who withdrew before participating (i.e., those who do not fill out any daily or weekly surveys), or discontinued the intervention (withdraw with less than 8 weeks of participation). The 'per protocol' cohort will include those who completed at least 8 weeks of study. The investigators define, for each participant, the amount of time that participants participated as the difference between the clinic activation date and latest of either the automatically-generated time-stamp of the last completed daily or weekly survey or the collection date of the last swab, with a maximum of 12 weeks. Those who participated for at least 8 weeks (56 days) according to this calculation will be included in the 'per protocol' cohort. For analyses using person time, the investigators will use the latest of the following; the last survey completed date or collection date from a swab collection.

Decision Algorithm for serological influenza outcome adjudication:

This decision algorithm documents the process for which ResPECT participants will be determined to have had laboratory-confirmed influenza based on serological testing only. The possible outcomes are: laboratory confirmed influenza confirmed by serology (LCI-S) and no laboratory confirmed influenza event confirmed by serology (no LCI-S). In some cases, outcomes (either LCI-S or no LCI-S) will be imputed. The algorithm to classify and/or impute these outcomes is as follows:

Step 1: Determine Study Completion Determine if participants have completed the study (and thus in the 'per protocol' cohort) or if participants have not and thus are in the ITT cohort

Step 2: Determine serological influenza outcome for those in the 'per protocol' cohort 2a. For those individuals in the 'per protocol' cohort who have two serological samples, collected at the beginning and end of the season according to protocol, and who experience a four-fold rise in influenza hemagglutination inhibition antibody (HAI) titer to exactly 0 strains, classify the serological influenza outcome as no LCI-S.

2b. For those individuals in the 'per protocol' cohort who have two serological samples, collected at the beginning and end of the season according to protocol, and who experience a four-fold rise in influenza HAI antibody titer to one or more strains, classify the serological influenza outcome as LCI-S.

2c. For those individuals in the 'per protocol' cohort who do not have two serological samples, collected at the beginning and end of the season according to protocol or who are missing vaccination info or were vaccinated during the study, impute the serological influenza outcome as LCI-S. Missing LCI-S status will be imputed using standard multiple imputation techniques, creating multiple imputed datasets with no missing values for each analysis.

Step 3: Impute the LCI-S outcome for the ITT cohort Some members of the ITT cohort did not complete all weeks of the study and may be missing a serological outcome for the same reasons mentioned above. For these individuals, the serological influenza outcome must be imputed. Missing LCI-S status will be imputed using standard multiple imputation techniques, creating multiple imputed datasets with no missing values for each analysis.

2.d Model and variable selection

This data is from a cluster-randomized clinical trial. The investigators anticipate that the constrained randomization will ensure balance across important covariates. The clinics were pair-matched by the following characteristics:

Study site Clinic size Clinic type (ED/Urgent care, Primary Care, Outpatient, Enhanced) Enhanced PPE (whether HCWs wore enhanced PPE during patient procedures, e.g. in dental and dialysis clinics) Patient population (Pediatric, Adult, or mixed)

Because these variables were matched on, the investigators will not adjust for any of them in the multivariable regression models. However, cluster-level random intercepts as well as additional participant-level covariates will be added to the model to adjust for possible residual confounding that is not controlled for by the cluster-randomized design. These covariates will be individual-level variables including:

Age, Gender, Race (White, Black or African American, Asian, Native Hawaiian or Pacific Islander, American Indian or Alaskan Native) and ethnicity (Hispanic or Latino) Number of household members under 5 (this has been noted as a strong risk factor for influenza), Categorical occupation risk level (low, medium, or high), Binary season-specific flu vaccination status (was or was not vaccinated), Proportion of daily surveys where an individual reported exposure to someone with respiratory symptoms, and Individual-level (self-reported) measures of mask and hand hygiene compliance.

The investigators will attempt to include all of the above-listed variables in the analysis. No variable selection will be performed to optimize the goodness of fit of the model. No Type I error rate adjustments will be made. Variables will be left out only if the variable contribute to instability in model estimation: e.g. collinearity (identified by variance inflation factors) or insufficient data to impute covariate status. In the model design stage, the investigators identified a full set of covariates that would satisfy the sample size recommendation that the investigators have no more than m/15 parameters in the model, where m = min(n1, n2) and n1 and n2 are the numbers in each of the response variable categories. Based on preliminary estimates of the total number of influenza outcomes expected, the investigators aimed to keep the number of estimated parameters below 25.

The following variables were considered but not included in the analysis for the final model. Justification is provided.

Follow-up variables such as contact with household members with flu: noisy, lacking flu confirmation, and too reliant on self-reporting biases.

Cumulative study-based vaccination status (i.e. ever vaccinated, never vaccinated): would be collinear with seasonal vaccine status.

Absence from work: not directly related to outcome, chose to include average number of hours worked instead.

Dummy variables of clinic types: while these encode important questions, they aren't the main purpose of the central study, and were characteristics that were matched on.

Size of household: for parsimony, the investigators will include number of household members under 5 instead.

Clinic size: was used in matching for randomization. Comorbid conditions: hard to justify including some and not others, of secondary relevance to the main outcome.

Average number of hours worked per week defined each season for each individual: there was a minimum number of hours worked defined in inclusion criteria, so this range will not be substantial.

Smoking status: secondary relevance to main outcome.

2.e Pre-specified exploratory analyses In addition to the pre-specified analyses of primary and secondary outcomes, the investigators will run several pre-specified exploratory analyses to assess the impact of vaccine coverage and protocol compliance with the study outcomes.

Using the models described in Sections 3 and 4 below, the investigators will consider adding additional covariates to the models from the primary and secondary analyses. Specifically, the investigators will examine the impact of covariates specific to a particular cluster-season including:

Vaccine coverage among participants in the cluster Hand-hygiene compliance rate Measure of how often any HCW in the clinic wore any mask, MM or N95 Proportion of clinic HCW enrolled in study and size of clinic

Additionally, the investigators will assess interaction terms considering the following variables:

Interaction of cluster-level mask compliance with mask group Interaction of individual-level vaccination status with mask group

Finally, the investigators will investigate combinations of cluster-level, seasonal, individual-level and cluster-seasonal random effects to capture different possible correlation structures of the data. The magnitude of each variance component will dictate whether the variance components are included in the final model.

3. Analysis plan for primary outcome: laboratory-confirmed influenza

3.a Outcome definitions A dichotomous variable will indicate whether or not a participant had an episode of laboratory-confirmed influenza during a single influenza season. As specified in the protocol, individuals who have a PCR-confirmed influenza infection collected within seven days of symptom onset or who have a 4-fold rise in antibody titer will be considered as a positive case, As described above, the investigators will implement a per-protocol analysis and an ITT analysis.

3.b Planned descriptive analysis The descriptive analysis will focus on aggregated participant numbers across the groups specified in "respect outcome tables.xlsx". The tables are as follows: 1) demographics, comprised of a breakout across treatment arms of characteristics including age, race, gender, occupation, clinic characteristics, vaccination status, and comorbid conditions, 2) Adjudication, where tallies of ResPECT participants are broken down into categories depending on participant's eligibility for the ITT and PP analyses and influenza adjudication outcome by year, 3) Nasopharyngeal swab lab results, where participants are broken out by year and mask type across the possible influenza and non-influenza viruses tested during the study, and 4) Summary results of lab-confirmed influenza, lab-confirmed non-influenza, ARI, LCRI, LDRI and ILI across intervention arms only.

3.c Planned Primary Analysis The investigators will use an individual-level logistic regression model to estimate the difference in influenza infection between the N95 and medical mask groups. Let Y_ijs be an indicator of whether subject i in cluster j developed laboratory-confirmed influenza in season s, and MASK_js is an indicator of which mask the clinic was assigned to in season s (0 if medical mask and 1 if N95). Then the investigators will fit a version of this model logit[Pr(Y_{ijs}=1|MASK_{js})]=Beta_{0}+Beta_{1}*MASK_{js}+SUM_{k}(Theta_{k}*X_{k,ijs}+alpha_{j} + alpha_{i} where the alpha_{j} are the cluster-level random intercepts, the alpha_{i} are the individual-level random intercepts (both assumed to be normally distributed), and the X_{k} refer to the individual-level covariates listed in Section 2.d. Unadjusted analyses will drop individual-level covariates and random intercepts, but will retain the cluster-level random effects.

For each fitted model, the estimated odds ratio comparing the odds of infection for those HCPs wearing N95s compared to those HCPs wearing medical masks (i.e. exp(Beta_{1}) will be reported, with a 95% confidence interval (CI).

The ITT and PP will use the same model equation (shown above) but will use different subsets of participants from the full cohort as described above.

3.d Planned Sensitivity Analysis To account for the unavoidable additional uncertainty regarding the missing data from the primary outcome, the investigators will conduct a sensitivity analysis that randomly assigns binary outcomes to participants who did not complete the study. Specifically, the investigators will create a two-dimensional grid on which the investigators vary the influenza attack rates in participants who dropped out of the study for both the medical mask (MM) and N95 arm, separately. The investigators will fix the MM dropout attack rate between half and twice the observed MM attack rate, based on complete data. The investigators will fix the N95 dropout attack rate between half and twice the observed N95 attack rate, based on complete data. By varying these two parameters across the grid, and for each combination, calculating the adjusted odds ratio (averaged across n=50 imputed datasets for each point on the grid), the investigators will observe the sensitivity of the results to values of the missing data.

Additionally, the investigators will compare rates reporting of symptomatic events in the two study arms. If the investigators detect a statistically significant difference in symptomatic reporting between arms, the investigators will include a covariate adjustment of person time in each model to account for the amount of person time under observation.

4. Analysis plan for secondary outcomes

4.a Definitions of secondary outcomes: Acute Respiratory Illness (ARI): This outcome is the incidence of ARI as a clinical syndrome. ARI will be defined as the occurrence of signs or symptoms of respiratory infection, as defined by Table 2 in the published protocol with or without laboratory confirmation.

Influenza-Like Illness (ILI): This outcome is the incidence of ILI as a clinical syndrome. ILI will be defined as temperature of 100°F [37.8°C] or greater plus cough and/or a sore throat, with or without laboratory confirmation.

Laboratory Confirmed Respiratory Illness (LCRI): This outcome is defined as a laboratory confirmed respiratory illness from any of the pathogens listed in Table 4 in the protocol. Laboratory confirmed respiratory illness is ARI combined with laboratory confirmation by reverse transcription-polymerase chain reaction (RT-PCR) of infection with any of the pathogens listed in Table 4 in an upper respiratory specimen swab after symptoms were reported and within seven days of the original symptomatic report (PP definition of LCRI and confirmed April, 2016). Events with multiple viruses detected will count as a single event of LCRI. If a swab that tested positive but was not associated with a symptomatic event (i.e. was not collected between symptom onset and seven days after symptom onset) then the incident does not count as a LCRI event. If an individual seroconverts to influenza, had symptoms at some time during the study, and does not have a PCR-confirmed pathogen event already, then the investigators will assign them a single LCRI event.

Laboratory-detected respiratory infection (LDRI): For a participant with or without symptoms, a laboratory-detected infection is defined as: 1) detection of a respiratory pathogen by PCR or other laboratory methods or 2) serological evidence of infection (e.g., seroconversion) with a respiratory pathogen during the study surveillance period(s). In a case where two or more pathogens are identified in the same specimen, each pathogen will be considered to represent a separate infection (e.g., 2 pathogens as 2 events, 3 pathogens as 3 events) for that study participant for that time-point. Sequential detection of the same pathogens by PCR or other laboratory method in swabs collected at least 21 days apart will be considered separate infections.

For all of these endpoints, an individual may experience any or all of the outcomes more than once during the course of the 12-week study. Within the same study identification (ID), participants must report being symptom-free for at least seven days prior to the beginning of the second event, except for LDRI which has the longer 21-day window separating events. As in the primary endpoint section, the secondary outcomes analysis will also include a per-protocol and an ITT analysis. A general description of these approaches is provided above, with specific modifications discussed below.

4.b Planned secondary outcome ITT analysis As in the primary outcome ITT, this analysis will include all of the randomized ResPECT participants regardless of withdrawal status, participation, or protocol adherence. Secondary outcomes will be characterized using a per-week rate of infection so that all participants may be included. The investigators will use a covariate-adjusted individual-level log-linear Poisson regression analysis with person time as an offset term as well as cluster-level and individual-level random intercepts. For the ITT analysis, the amount of person time will be fixed at 12 weeks for each participant, regardless of how much time participant participated in the study. The investigators will include the same covariates as described in the primary outcome analysis section above in the Poisson regression model for the ITT and per-protocol analyses. Unadjusted models will include only the cluster-level random intercepts.

For each fitted model, the estimated incidence rate ratio between the N95 and medical mask arm will be estimated and reported, with a 95% CI.

4.c Secondary outcome per-protocol analysis Per-protocol analyses will use the same Poisson regression methods described for the secondary outcome ITT analyses. Additionally, the per-protocol analyses will include ResPECT study participants who completed at least 8 weeks (starting at the time of site activation) of the 12-week trial. All randomized participants will be included unless participant withdrew, were administratively withdrawn, or deactivated before participating for at least 8 weeks.

Calculation of person-weeks for each participant will proceed as follows: for individuals who withdrew, completion date will be determined by the earliest withdrawal or deactivation date; in the event that these dates conflict, the earlier date will be used. For all other participants, active participation time will be calculated as the time between clinic activation and the latest of either the automatically-generated timestamp of the last completed daily or weekly survey or the collection date of the last swab, up to 12 weeks.

4.d Missing covariate data for secondary outcomes The analysis approaches for the secondary outcomes will encounter instances of missing data, either in or failure to report relevant information on self-reported forms. Areas in which these issues may require special handling are 1) missing swab collection dates, 2) missing swab results, and 3) incomplete symptomatic event reporting.

Missing swab collection dates are relevant for matching swab results to symptomatic event reports. Where this data is missing (often in the case of swabs collected using take-home kits, where participants self-collected the nasopharyngeal (NP) samples), the investigators will attempt to match swab results to symptomatic reporting events using the swab number or process of elimination (ie, only one event was reported and only 1 symptomatic swab was provided).

Missing swab results may occur due to practical considerations (running out of PCR plates), participant noncompliance, or handling errors. These results are truly missing, cannot be recovered, and therefore must be discarded. There are also a few instances (<30 out of >11,000, or <0.27%) in which results cannot be reliably matched to the correct individual due to barcode transcription errors. These will be discarded if there is any doubt about the correct assignment barcode. Since these errors did not arise in a systematic way and comprise a very small portion of the overall available and reliable swab samples, this decision should not affect the analysis outcome.

A few instances also exist in which participants provided a symptomatic swab but failed to complete a symptomatic event form. Since the participant provided no details to accompany the biological specimen, the investigators will not include these data in the analysis of ILI events (which require specific symptom reports). However, positive symptomatic swab data lacking specific symptom data will be included in the ARI and LCRI.

ELIGIBILITY:
Inclusion Criteria:

* Clinical site leadership has agreed to have one or more staff participate in the trial
* Subject meets the definition of "healthcare personnel"
* Subject able to read and sign informed consent
* Subject agrees to all requirements of the protocol, including fit testing and diary keeping
* Subject's age is 18 or greater
* Subject passes fit testing for one of the study supplied respirator models and agrees to use that model for the entire intervention period of the study (if in respirator arm).

Exclusion Criteria:

* Subject self-identified as having severe heart, lung, neurological or other systemic disease that one or more Investigator believes could preclude safe participation
* Known to not tolerate wearing respiratory protective equipment for any period
* Facial hair, or other issue such as facial adornments, precluding respirator OSHA-compliant fit testing or proper mask fit during the study period
* Advised by Occupational Health (or other qualified clinician) to not wear the same or similar respirator or medical mask models used in this study
* In the opinion of the Investigator, may not be able to reasonably participate in the trial for any reason
* Self-identified as in, or will be in the third trimester of pregnancy, during the study period.
* Subject rotating in 2 different ResPECT study clinic sites /clusters during the 12-week study period.
* Subject works less than 75% of the intervention period in that clinic.
* Subject is a previous participant of the ResPECT Study, but does not consent for data from previous flu season(s) to be linked.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2862 (Actual)
Dates: Start 2010-12; Primary Completion 2018-03 (Actual); Study Completion 2018-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Trish M. Perl, MD, Principal Investigator — UTSouthwestern Medical Center; Lewis Radonovich, MD, Principal Investigator — CDC-NIOSH; Derek Cummings, PhD, Study Director — University of Florida; Michael Simberkoff, MD, Study Director — New York Harbor Healthcare System VA; Connie S Price, MD, Study Director — University of Colorado (Denver Health); Charlotte Gaydos, PhD, Study Director — Johns Hopkins University; Nicholas Reich, PhD, Study Director — University of Massachusetts, Amherst
Locations (7):
- United States (7):
  - Children's Hospital Colorado Infectious Disease, Aurora, Colorado
  - Denver Health Medical Center, Denver, Colorado
  - Denver Veteran's Administration Medical Center, Denver, Colorado
  - Veterans Affairs Medical Center, Washington, DC, Washington D.C., District of Columbia
  - Johns Hopkins Health Sytstem, Baltimore, Maryland
  - VA New York Harbor Healthcare System, New York, New York
  - Houston VA Medical Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anzueto A, Niederman MS. Diagnosis and treatment of rhinovirus respiratory infections. Chest. 2003 May;123(5):1664-72. doi: 10.1378/chest.123.5.1664. PMID 12740288
- [Background] Askarian M, Mirzaei K, Honarvar B, Etminan M, Araujo MW. Knowledge, attitude and practice towards droplet and airborne isolation precautions among dental health care professionals in Shiraz, Iran. J Public Health Dent. 2005 Winter;65(1):43-7. doi: 10.1111/j.1752-7325.2005.tb02785.x. PMID 15751494
- [Background] Askarian M, Mirzaei K, Mundy LM, McLaws ML. Assessment of knowledge, attitudes, and practices regarding isolation precautions among Iranian healthcare workers. Infect Control Hosp Epidemiol. 2005 Jan;26(1):105-8. doi: 10.1086/502495. PMID 15693417
- [Background] Bettinardi O, Argentero P, Giorgi I. [Assessment of occupational stress among workers in rehabilitation medicine]. G Ital Med Lav Ergon. 2007 Jul-Sep;29(3 Suppl):693-5. Italian. PMID 18409908
- [Background] Blachere FM, Lindsley WG, Pearce TA, Anderson SE, Fisher M, Khakoo R, Meade BJ, Lander O, Davis S, Thewlis RE, Celik I, Chen BT, Beezhold DH. Measurement of airborne influenza virus in a hospital emergency department. Clin Infect Dis. 2009 Feb 15;48(4):438-40. doi: 10.1086/596478. PMID 19133798
- [Background] Bly JL. Measuring productivity for home health nurses. Home Health Care Serv Q. 1981 Fall;2(3):23-39. doi: 10.1300/j027v02n03_03. PMID 10255198
- [Background] Booth TF, Kournikakis B, Bastien N, Ho J, Kobasa D, Stadnyk L, Li Y, Spence M, Paton S, Henry B, Mederski B, White D, Low DE, McGeer A, Simor A, Vearncombe M, Downey J, Jamieson FB, Tang P, Plummer F. Detection of airborne severe acute respiratory syndrome (SARS) coronavirus and environmental contamination in SARS outbreak units. J Infect Dis. 2005 May 1;191(9):1472-7. doi: 10.1086/429634. Epub 2005 Mar 18. PMID 15809906
- [Background] Brankston G, Gitterman L, Hirji Z, Lemieux C, Gardam M. Transmission of influenza A in human beings. Lancet Infect Dis. 2007 Apr;7(4):257-65. doi: 10.1016/S1473-3099(07)70029-4. PMID 17376383
- [Background] Bridges CB, Kuehnert MJ, Hall CB. Transmission of influenza: implications for control in health care settings. Clin Infect Dis. 2003 Oct 15;37(8):1094-101. doi: 10.1086/378292. Epub 2003 Sep 19. PMID 14523774
- [Background] Burke JP. Infection control - a problem for patient safety. N Engl J Med. 2003 Feb 13;348(7):651-6. doi: 10.1056/NEJMhpr020557. No abstract available. PMID 12584377
- [Background] Cadena J, Thompson GR 3rd, Patterson JE, Nakashima B, Owens A, Echevarria K, Mortensen EM. Clinical predictors and risk factors for relapsing Clostridium difficile infection. Am J Med Sci. 2010 Apr;339(4):350-5. doi: 10.1097/MAJ.0b013e3181d3cdaa. PMID 20224312
- [Background] Chia SE, Koh D, Fones C, Qian F, Ng V, Tan BH, Wong KS, Chew WM, Tang HK, Ng W, Muttakin Z, Emmanuel S, Fong NP, Koh G, Lim MK. Appropriate use of personal protective equipment among healthcare workers in public sector hospitals and primary healthcare polyclinics during the SARS outbreak in Singapore. Occup Environ Med. 2005 Jul;62(7):473-7. doi: 10.1136/oem.2004.015024. PMID 15961624
- [Background] Chor JS, Ngai KL, Goggins WB, Wong MC, Wong SY, Lee N, Leung TF, Rainer TH, Griffiths S, Chan PK. Willingness of Hong Kong healthcare workers to accept pre-pandemic influenza vaccination at different WHO alert levels: two questionnaire surveys. BMJ. 2009 Aug 25;339:b3391. doi: 10.1136/bmj.b3391. PMID 19706937
- [Background] Christini AB, Shutt KA, Byers KE. Influenza vaccination rates and motivators among healthcare worker groups. Infect Control Hosp Epidemiol. 2007 Feb;28(2):171-7. doi: 10.1086/511796. Epub 2007 Jan 17. PMID 17265398
- [Background] Daley P, Castriciano S, Chernesky M, Smieja M. Comparison of flocked and rayon swabs for collection of respiratory epithelial cells from uninfected volunteers and symptomatic patients. J Clin Microbiol. 2006 Jun;44(6):2265-7. doi: 10.1128/JCM.02055-05. PMID 16757636
- [Background] Daugherty EL, Perl TM, Needham DM, Rubinson L, Bilderback A, Rand CS. The use of personal protective equipment for control of influenza among critical care clinicians: A survey study. Crit Care Med. 2009 Apr;37(4):1210-6. doi: 10.1097/CCM.0b013e31819d67b5. PMID 19242326
- [Background] Daugherty EL, Perl TM, Rubinson L, Bilderback A, Rand CS. Survey study of the knowledge, attitudes, and expected behaviors of critical care clinicians regarding an influenza pandemic. Infect Control Hosp Epidemiol. 2009 Dec;30(12):1143-9. doi: 10.1086/648085. PMID 19877816
- [Background] de Gentile A, Rivas N, Sinkowitz-Cochran RL, Momesso T, Iriart EM, Lopez E, Beck-Sague CM, Jarvis WR. Nosocomial infections in a children's hospital in Argentina: impact of a unique infection control intervention program. Infect Control Hosp Epidemiol. 2001 Dec;22(12):762-6. doi: 10.1086/501859. PMID 11876454
- [Background] Drinka PJ, Gravenstein S, Krause P, Langer EH, Barthels L, Dissing M, Shult P, Schilling M. Non-influenza respiratory viruses may overlap and obscure influenza activity. J Am Geriatr Soc. 1999 Sep;47(9):1087-93. doi: 10.1111/j.1532-5415.1999.tb05232.x. PMID 10484251
- [Background] Dudukgian H, Sie E, Gonzalez-Ruiz C, Etzioni DA, Kaiser AM. C. difficile colitis--predictors of fatal outcome. J Gastrointest Surg. 2010 Feb;14(2):315-22. doi: 10.1007/s11605-009-1093-2. PMID 19937192
- [Background] Elder AG, O'Donnell B, McCruden EA, Symington IS, Carman WF. Incidence and recall of influenza in a cohort of Glasgow healthcare workers during the 1993-4 epidemic: results of serum testing and questionnaire. BMJ. 1996 Nov 16;313(7067):1241-2. doi: 10.1136/bmj.313.7067.1241. No abstract available. PMID 8939114
- [Background] Evans ME, Hall KL, Berry SE. Influenza control in acute care hospitals. Am J Infect Control. 1997 Aug;25(4):357-62. doi: 10.1016/s0196-6553(97)90029-8. PMID 9276549
- [Background] Fendrick AM, Monto AS, Nightengale B, Sarnes M. The economic burden of non-influenza-related viral respiratory tract infection in the United States. Arch Intern Med. 2003 Feb 24;163(4):487-94. doi: 10.1001/archinte.163.4.487. PMID 12588210
- [Background] Ferguson NM, Cummings DA, Fraser C, Cajka JC, Cooley PC, Burke DS. Strategies for mitigating an influenza pandemic. Nature. 2006 Jul 27;442(7101):448-52. doi: 10.1038/nature04795. Epub 2006 Apr 26. PMID 16642006
- [Background] Fisher E, Rengasamy S, Viscusi D, Vo E, Shaffer R. Development of a test system to apply virus-containing particles to filtering facepiece respirators for the evaluation of decontamination procedures. Appl Environ Microbiol. 2009 Mar;75(6):1500-7. doi: 10.1128/AEM.01653-08. Epub 2009 Jan 9. PMID 19139225
- [Background] Gammon J, Morgan-Samuel H, Gould D. A review of the evidence for suboptimal compliance of healthcare practitioners to standard/universal infection control precautions. J Clin Nurs. 2008 Jan;17(2):157-67. doi: 10.1111/j.1365-2702.2006.01852.x. Epub 2007 Mar 1. PMID 17331098
- [Background] Gershon RR, Karkashian CD, Vlahov D, Kummer L, Kasting C, Green-McKenzie J, Escamilla-Cejudo JA, Kendig N, Swetz A, Martin L. Compliance with universal precautions in correctional health care facilities. J Occup Environ Med. 1999 Mar;41(3):181-9. doi: 10.1097/00043764-199903000-00007. PMID 10091141
- [Background] Ginocchio CC. Detection of respiratory viruses using non-molecular based methods. J Clin Virol. 2007 Nov;40 Suppl 1:S11-4. doi: 10.1016/S1386-6532(07)70004-5. PMID 18162248
- [Background] Grinshpun SA, Haruta H, Eninger RM, Reponen T, McKay RT, Lee SA. Performance of an N95 filtering facepiece particulate respirator and a surgical mask during human breathing: two pathways for particle penetration. J Occup Environ Hyg. 2009 Oct;6(10):593-603. doi: 10.1080/15459620903120086. PMID 19598054
- [Background] Jarvis WR. Infection control and changing health-care delivery systems. Emerg Infect Dis. 2001 Mar-Apr;7(2):170-3. doi: 10.3201/eid0702.010202. PMID 11294699
- [Background] Jefferson T, Foxlee R, Del Mar C, Dooley L, Ferroni E, Hewak B, Prabhala A, Nair S, Rivetti A. Physical interventions to interrupt or reduce the spread of respiratory viruses: systematic review. BMJ. 2008 Jan 12;336(7635):77-80. doi: 10.1136/bmj.39393.510347.BE. Epub 2007 Nov 27. PMID 18042961
- [Background] Johnson DF, Druce JD, Birch C, Grayson ML. A quantitative assessment of the efficacy of surgical and N95 masks to filter influenza virus in patients with acute influenza infection. Clin Infect Dis. 2009 Jul 15;49(2):275-7. doi: 10.1086/600041. PMID 19522650
- [Background] Loeb M, Dafoe N, Mahony J, John M, Sarabia A, Glavin V, Webby R, Smieja M, Earn DJ, Chong S, Webb A, Walter SD. Surgical mask vs N95 respirator for preventing influenza among health care workers: a randomized trial. JAMA. 2009 Nov 4;302(17):1865-71. doi: 10.1001/jama.2009.1466. Epub 2009 Oct 1. PMID 19797474
- [Background] Radonovich LJ Jr, Cheng J, Shenal BV, Hodgson M, Bender BS. Respirator tolerance in health care workers. JAMA. 2009 Jan 7;301(1):36-8. doi: 10.1001/jama.2008.894. No abstract available. PMID 19126810
- [Background] Radonovich LJ Jr, Hodgson MJ, Cohen HJ. Do respirators protect health-care workers from airborne infectious diseases? Respir Care. 2008 Dec;53(12):1660-4. No abstract available. PMID 19025698
- [Background] Radonovich LJ Jr, Perl TM, Davey V, Cohen H. Preventing the soldiers of health care from becoming victims on the pandemic battlefield: respirators or surgical masks as the armor of choice. Disaster Med Public Health Prep. 2009 Dec;3 Suppl 2:S203-10. doi: 10.1097/DMP.0b013e3181be830c. PMID 19794307
- [Background] Rengasamy S, Eimer BC, Shaffer RE. Comparison of nanoparticle filtration performance of NIOSH-approved and CE-marked particulate filtering facepiece respirators. Ann Occup Hyg. 2009 Mar;53(2):117-28. doi: 10.1093/annhyg/men086. PMID 19261695
- [Background] Whitehead J. Sample size calculations for ordered categorical data. Stat Med. 1993 Dec 30;12(24):2257-71. doi: 10.1002/sim.4780122404. PMID 8134732
- [Background] Radonovich LJ Jr, Bessesen MT, Cummings DA, Eagan A, Gaydos C, Gibert C, Gorse GJ, Nyquist AC, Reich NG, Rodrigues-Barradas M, Savor-Price C, Shaffer RE, Simberkoff MS, Perl TM. The Respiratory Protection Effectiveness Clinical Trial (ResPECT): a cluster-randomized comparison of respirator and medical mask effectiveness against respiratory infections in healthcare personnel. BMC Infect Dis. 2016 Jun 2;16:243. doi: 10.1186/s12879-016-1494-2. PMID 27255755
- [Background] Schafer JL. Multiple imputation: a primer. Stat Methods Med Res. 1999 Mar;8(1):3-15. doi: 10.1177/096228029900800102. PMID 10347857
- [Background] Williams CJ, Schweiger B, Diner G, Gerlach F, Haaman F, Krause G, Nienhaus A, Buchholz U. Seasonal influenza risk in hospital healthcare workers is more strongly associated with household than occupational exposures: results from a prospective cohort study in Berlin, Germany, 2006/07. BMC Infect Dis. 2010 Jan 12;10:8. doi: 10.1186/1471-2334-10-8. PMID 20067628
- [Background] U.S. Department of Health and Human Services: Food and Drug Administration (2005). Guidance for Industry: Collection of Race and Ethnicity Data in Clinical Trials. Rockville, MD: Food and Drug Administration.
- [Background] Fisher LD, Dixon DO, Herson J, et al. (1990) Intention to treat in clinical trials. In: Peace KE (Ed.), Statistical issues in drug research and development (pp. 331-50). New York, NY: Marcel Dekker.
- [Background] Hayes RJ and Moulton LH (2009) Cluster Randomised Trials. Chapman and Hall/CRC.
- [Background] ICH Expert Working Group (1998). ICH Harmonised Tripartite Guideline, Statistical Principles for Clinical Trials E9, Current Step 4 version dated 5 February 1998. http://www.ich.org/fileadmin/Public_Web_Site/ICH_Products/Guidelines/Efficacy/E9/Step4/E9_Guideline.pdf (last accessed 04 June 2017).
- [Derived] Jefferson T, Dooley L, Ferroni E, Al-Ansary LA, van Driel ML, Bawazeer GA, Jones MA, Hoffmann TC, Clark J, Beller EM, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2023 Jan 30;1(1):CD006207. doi: 10.1002/14651858.CD006207.pub6. PMID 36715243
- [Derived] Los J, Gaydos CA, Gibert CL, Gorse GJ, Lykken J, Nyquist AC, Price CS, Radonovich LJ Jr, Rattigan S, Reich N, Rodriguez-Barradas M, Simberkoff M, Bessesen M, Brown A, Cummings DAT, Perl TM; ResPECT Study Team. Take-home kits to detect respiratory viruses among healthcare personnel: Lessons learned from a cluster randomized clinical trial. Am J Infect Control. 2021 Jul;49(7):893-899. doi: 10.1016/j.ajic.2021.02.001. Epub 2021 Feb 10. PMID 33581146
- [Derived] Jefferson T, Del Mar CB, Dooley L, Ferroni E, Al-Ansary LA, Bawazeer GA, van Driel ML, Jones MA, Thorning S, Beller EM, Clark J, Hoffmann TC, Glasziou PP, Conly JM. Physical interventions to interrupt or reduce the spread of respiratory viruses. Cochrane Database Syst Rev. 2020 Nov 20;11(11):CD006207. doi: 10.1002/14651858.CD006207.pub5. PMID 33215698
- [Derived] Cummings DAT, Radonovich LJ, Gorse GJ, Gaydos CA, Bessesen MT, Brown AC, Gibert CL, Hitchings MDT, Lessler J, Nyquist AC, Rattigan SM, Rodriguez-Barradas MC, Price CS, Reich NG, Simberkoff MS, Perl TM. Risk Factors for Healthcare Personnel Infection With Endemic Coronaviruses (HKU1, OC43, NL63, 229E): Results from the Respiratory Protection Effectiveness Clinical Trial (ResPECT). Clin Infect Dis. 2021 Dec 6;73(11):e4428-e4432. doi: 10.1093/cid/ciaa900. PMID 32645144
- [Derived] Radonovich LJ Jr, Simberkoff MS, Bessesen MT, Brown AC, Cummings DAT, Gaydos CA, Los JG, Krosche AE, Gibert CL, Gorse GJ, Nyquist AC, Reich NG, Rodriguez-Barradas MC, Price CS, Perl TM; ResPECT investigators. N95 Respirators vs Medical Masks for Preventing Influenza Among Health Care Personnel: A Randomized Clinical Trial. JAMA. 2019 Sep 3;322(9):824-833. doi: 10.1001/jama.2019.11645. PMID 31479137
- [Derived] Lauer SA, Kleinman KP, Reich NG. The effect of cluster size variability on statistical power in cluster-randomized trials. PLoS One. 2015 Apr 1;10(4):e0119074. doi: 10.1371/journal.pone.0119074. eCollection 2015. PMID 25830416
- [Derived] Reich NG, Myers JA, Obeng D, Milstone AM, Perl TM. Empirical power and sample size calculations for cluster-randomized and cluster-randomized crossover studies. PLoS One. 2012;7(4):e35564. doi: 10.1371/journal.pone.0035564. Epub 2012 Apr 27. PMID 22558168
- See also: The National Institute for Occupational Safety and Health (NIOSH) — http://www.cdc.gov/niosh/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: participants were recruited from outpatient settings considered at high risk for respiratory illnesses (emergency rooms, internal medicine and pediatric clinics) and had to work at least 24 hours per week in a given setting. They had to have face to face exposure to patients and be willing and able to participate, sign informed consent.
Groups:
- N95 Respirator: The investigators are comparing the selected N95 respirators against the selected medical mask.
  N95 Respirator: Participants in this arm will be asked to wear an N95 respirator for the extent of the 12 week study period.
- Medical/Surgical Mask: The investigators are comparing the selected medical/surgical mask against the N95 respirator.
  Medical/surgical mask: Participants in this arm will be asked to wear a medical/surgical mask for the extent of the 12 week study period.
Period: Overall Study
Arm/Group | N95 Respirator | Medical/Surgical Mask
Started | 1374 | 1488
Completed | 1374 | 1488
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | N95 Respirator | Medical/Surgical Mask | Total
Number analyzed (Participants) | 1374 | 1488 | 2862
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1347 | 1451 | 2798
  >=65 years | 27 | 37 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (0.6) | 43 (0.5) | 43 (0.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1149 | 1220 | 2369
  Male | 225 | 268 | 493
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 212 | 227 | 439
  Not Hispanic or Latino | 1151 | 1245 | 2396
  Unknown or Not Reported | 11 | 16 | 27
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 9 | 7 | 16
  Asian | 103 | 108 | 211
  Native Hawaiian or Other Pacific Islander | 2 | 6 | 8
  Black or African American | 371 | 431 | 802
  White | 731 | 761 | 1492
  More than one race | 50 | 57 | 107
  Unknown or Not Reported | 108 | 118 | 226
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1374 | 1488 | 2862

OUTCOME MEASURES:

1. Primary Outcome: Protective Effects of N95 Respirators vs Medical Masks (MM) as Assessed by Number of Influenza A and B Events
Description: Number of influenza A and B events in healthcare practitioners wearing N95 respirators compared to medical masks.
Time Frame: 60 weeks
Measure: Number; unit: number of influenza A and B events
Arm/Group | N95 Respirator | Medical/Surgical Mask
Number analyzed (Participants) | 1374 | 1488
number of influenza A and B events | 222 | 204

2. Secondary Outcome: Protective Effects of N95 Respirators vs Medical Masks as Assessed by Number of Influenza-like Illnesses
Description: Number of influenza-like illnesses in healthcare practitioners wearing N95 respirators compared to medical masks.
Time Frame: 60 weeks
Measure: Number; unit: number of influenza-like illnesses
Arm/Group | N95 Respirator | Medical/Surgical Mask
Number analyzed (Participants) | 1374 | 1488
number of influenza-like illnesses | 128 | 166

3. Secondary Outcome: Protective Effects of N95 Respirators vs Medical Masks as Assessed by Number of Lab Confirmed Respiratory Illnesses
Description: Number of lab confirmed respiratory illnesses in healthcare practitioners wearing N95 respirators compared to medical masks.
Time Frame: 60 weeks
Measure: Number; unit: number of respiratory illnesses
Arm/Group | N95 Respirator | Medical/Surgical Mask
Number analyzed (Participants) | 1374 | 1488
number of respiratory illnesses | 371 | 417

4. Secondary Outcome: Protective Effects of N95 Respirators vs Medical Masks as Assessed by Number of Lab Detected Respiratory Infections
Description: Number of lab detected respiratory infections in healthcare practitioners wearing N95 respirators compared to medical masks.
Time Frame: 60 weeks
Measure: Number; unit: number of respiratory infections
Arm/Group | N95 Respirator | Medical/Surgical Mask
Number analyzed (Participants) | 1374 | 1488
number of respiratory infections | 679 | 745

5. Secondary Outcome: Protective Effects of N95 Respirators vs Medical Masks as Assessed by Number of Acute Respiratory Illnesses
Description: Number of acute respiratory illnesses in healthcare practitioners wearing N95 respirators compared to medical masks.
Time Frame: 60 weeks
Measure: Number; unit: number of acute respiratory illnesses
Arm/Group | N95 Respirator | Medical/Surgical Mask
Number analyzed (Participants) | 1374 | 1488
number of acute respiratory illnesses | 1556 | 1711

6. Secondary Outcome: Protective Effects of N95 Respirators vs Medical Masks as Assessed by Number of Laboratory Confirmed Illness
Description: Number of laboratory confirmed influenza illnesses in healthcare practitioners wearing N95 respirators compared to medical masks.
Time Frame: 60 weeks
Measure: Number; unit: Number of laboratory confirmed illnesses
Arm/Group | N95 Respirator | Medical/Surgical Mask
Number analyzed (Participants) | 1374 | 1488
Number of laboratory confirmed illnesses | 207 | 193

ADVERSE EVENTS:
Time Frame: We collected adverse events (AEs) for each 12-week respiratory season (total of 4 seasons) while participants were actively wearing masks or respirators.
Description: An AE is any adverse change from patient's baseline (pre-study) condition, which occurs during the course of the study, whether the event is considered to be related to the study intervention or not and documented in REDCap. Researchers assessed if the reported event meets the definition of an AE. Patients will be monitored until resolution. AEs were submitted to local Institutional Review Board according to their reporting policy. Participants reported symptoms in daily and weekly diaries.
Arm/Group | N95 Respirator | Medical/Surgical Mask
All-Cause Mortality (participants affected / at risk) | 0/1374 | 0/1488
Serious Adverse Events (participants affected / at risk) | 0/1374 | 0/1488
Other Adverse Events (participants affected / at risk) | 19/1374 | 0/1488
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | N95 Respirator (N=1374) | Medical/Surgical Mask (N=1488)
rash (Skin and subcutaneous tissue disorders) | 19 (19) | 0 (0) — skin irritation and worsening acne reported -- all events reported at one site in one respiratory virus season

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-17): https://cdn.clinicaltrials.gov/large-docs/25/NCT01249625/Prot_SAP_000.pdf